CLINICAL TRIAL: NCT03219242
Title: Longitudinal Prospective Study on Primary Debulking Surgery Including Bowel Resection in Advanced Stage Ovarian Cancer Patients Using Caiman® Technology
Brief Title: Primary Debulking Surgery Including Bowel Resection in Advanced Stage Ovarian Cancer Using Caiman® Technology
Acronym: CAIMAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Director, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25543/16
Record Dates: First submitted 2017-06-29; First posted 2017-07-17 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer
Keywords: Advanced ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Caiman device (Experimental): Time sparing and post-operative outcome in ovarian cancer including bowel resection for cytoreductive surgery with Caiman device
  Interventions: Device: Caiman® device

INTERVENTIONS:
Device: Caiman® device — Using CAIMAN device in primary surgery for ovarian cancer. Analyze potential time-sparing and the incidence of post-surgical complications.

SUMMARY:
Longitudinal prospective study on primary debulking surgery including bowel resection in advanced stage ovarian cancer patients using Caiman® technology

DETAILED DESCRIPTION:
Using CAIMAN® technology in primary surgery for advanced ovarian cancer including bowel resections.

Analyze potential time-sparing and the incidence of post-surgical complications.

Prospective, longitudinal, observational. 40 patients / year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years
* Patients with advanced ovarian cancer (FIGO stage IIIC-IV).
* Bowel resection
* Class 0-2 according to the American Society of Anesthesiologists (i.e.: ASA score ≤ 2)
* Written informed consent to the study

Exclusion Criteria:

* Pregnant or chronic infections
* Previous pelvic radiotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
time-sparing for bowel resection | up to 1 hour
  Time needed for bowel resection and radical omentecomy in avanced ovarian cancer
Post surgical complications | Up to 6 months
  F-up in 1-3 and 6 months with questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Professor, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart Rome,, Rome, Rome, Italy